CLINICAL TRIAL: NCT06082895
Title: The Effect of Motivational Interviewing Method on Birth Self-efficacy and Birth Satisfaction: A Randomized Controlled Study.
Brief Title: The Effect of Motivational Interviewing Method on Birth Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Sarı (Other)
Responsible Party: Sponsor-Investigator, Tuğba Sarı, sponsor-investigator, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TOGU-HEM-TS-02
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Self Efficacy
Keywords: birth self-efficacy; motivational interview; pregnancy

STUDY DESIGN:
Intervention Model Description: Two groups, intervention and control groups, will be created by randomization method for pregnant women who have fear of birth and are determined to have low birth self-efficacy. Pregnant women in the intervention group will be given a 4-session motivational interview program. The control group will continue routine monitoring. After the training, birth self-efficacy levels will be compared between the two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This group will consist of 45 pregnant women. The training program based on the motivational interviewing method will continue once a week for a total of 4 weeks.
  Interventions: Behavioral: Birth self-efficacy enhancement training based on motivational interviewing method
- control group (No Intervention): This group will consist of 45 pregnant women. This group will not be given any training program and routine pregnancy follow-ups will continue.

INTERVENTIONS:
Behavioral: Birth self-efficacy enhancement training based on motivational interviewing method — Birth self-efficacy enhancement training based on motivational interviewing method
  Arms: intervention group

SUMMARY:
Birth enables women to assume the role of parent, but experiencing labor pain is seen as a very stressful event. Birth pain is described as one of the most severe pains women experience throughout their lives. Different pharmacological and non-pharmacological methods are used to cope with labor pain. Non-pharmacological coping includes physiological coping (such as breathing techniques, relaxation, postural changes, and movement during labor), psychological coping (including social support, increasing self-efficacy, and increasing self-confidence), and cognitive coping (including distraction, illustration). , and focus). Birth self-efficacy refers to the mother's confidence or perception in her own ability to give birth, which may influence her future birth choices. Women with high efficacy expectations (i.e., high confidence regarding childbirth) may use cognitive coping behaviors to cope with labor pain and therefore reduce the likelihood of medical intervention.It has been found that a woman's confidence in her ability to cope with childbirth contributes significantly to her perception of pain during labor and can foster a positive perception of birth. Pregnant women with low self-efficacy also have low self-confidence during birth, which negatively affects their ability to take an active role during birth and causes an increase in cesarean delivery rates. Various approaches such as antenatal training, cognitive behavioral approach, and psychoeducation program are used to reduce the negative consequences that fear of birth may cause and to help pregnant women cope with the fear of birth and increase birth self-efficacy. One of the approaches that include these strategies is seen as the motivational interviewing method. The motivational interviewing method is a goal-oriented and more participant-centered counseling approach that aims to facilitate and activate participants' intrinsic motivation to change their behavior. Motivational interviewing is a method that encourages the participant to think about changes that can be made, rather than the counselor offering suggestions. The basic concepts of motivational interviewing are that the participant recognizes and accepts the need to make changes in their lives; This approach encourages participants to consider whether they are ready to change their behavior.

DETAILED DESCRIPTION:
Type of Research: The research will be conducted as a randomized controlled, experimental study to increase birth self-efficacy in pregnant women using the motivational interviewing method.

Population of the Research: The population of the research consists of pregnant women who came to the Gynecology and Obstetrics outpatient clinic between October 2023 and December 2023.

The sample of the Research G*Power version 3.1.9.7 program was used to calculate the research sample size and power value. It was calculated by taking a study as a reference in the sample size calculation. According to G power analysis, 5% margin of error, 95% power (representing the universe) and effect size were calculated as 70 in total, 35 in both groups. In the sample selection, pregnant women who have fear of childbirth and low self-efficacy will be selected as the main parameter of the study. In the literature review, it is seen that the fear of birth begins from the 20th week of pregnancy and increases throughout pregnancy. Therefore, pregnant women at or above the 20th week of pregnancy were included in the study. Pregnant women after 34 weeks were not included so that the training program was 4 weeks long and the participating pregnant women could complete the prenatal education. Taking into account the loss of pregnant women who met the research criteria and agreed to participate in the study, the sample size was determined as 90 participants, 45 for both groups. Creation of the Control and Experimental Group: After meeting the pregnant women who came for routine pregnancy examination and evaluating their suitability according to the research criteria, the Personal Information Form and the Short Version of the Self-Efficacy Scale in Labor were filled out by the pregnant women who met the inclusion criteria and volunteered to participate in the study. Pregnant women who had fear of childbirth and low self-efficacy were informed about the study and their written and verbal consent was obtained from the voluntary consent form. In addition, a list was prepared containing the name, surname, estimated date of birth based on the last menstrual period and contact information of the pregnant women.

Randomization Randomization technique was used to assign participants to groups. Stratification randomization technique will be used to ensure homogeneity according to the data obtained from the pregnant women (educational status, age and gestational week).

Blinding: Double blinding is not appropriate because the researcher included in the study provided training according to the motivational interviewing method, collected data on fear of birth, prenatal attachment and anxiety, and took part in the analysis of these data. However, pregnant women were assigned to the experimental and control groups by randomization, and one-sided blinding would be applied because the individuals did not interact with each other and did not know which group they were in.

Implementation of the Research The research was carried out in two separate stages. Stage 1: Preparatory phase Birth self-efficacy training program based on motivational interviewing method Phase 2: Implementation phase of the training program Preparation Process of the Training Program The first aim of the training program is to help women who are still pregnant cope with the fear of childbirth and low self-efficacy. For this purpose, studies and educational contents were examined to detect the negative emotional state caused by fear of birth and low self-efficacy and to develop positive emotional states. Specific to the motivational interviewing method in each session of the program; Open-ended questioning, reflective listening, confirmation and summarizing communication methods will be used. The first stage of motivational interviewing is to create internal motivation for change. In this direction; Session 1; Developing contradiction is an important method to reveal the talk of change in pregnant women. Conflict issues in pregnancy will be discussed by discussing the pregnant woman's thoughts, feelings, concerns, fears regarding birth and the effect of fear of birth on labor.

Session 2; In the first session, the interview will start with the homework given to the pregnant woman and the decision balance regarding the positive and negative characteristics of vaginal and cesarean birth. In this direction; Training will be given via computer slide presentation on the signs of labor onset, stages of labor, and cesarean delivery.

3rd Session; In order to evaluate the change process of the pregnant woman, her emotional state regarding the fear of birth will be reviewed and this issue will be discussed. A conflict will be created by evaluating the methods of coping with labor contractions and the level of knowledge about the birth environment.

4th Session; We will continue to develop a change plan and reveal commitment to strengthen commitment to change. The pregnant woman's birth-related goals are clarified and possible methods to achieve the chosen goals will be evaluated.

Implementation of the Experimental Group Training Program Within the scope of the research, pregnant women in the experimental group will be interviewed to determine the suitability of the place, time and hour of the training. After all pregnant women are interviewed and the appropriate time and day are determined for everyone, days when there is no training at the hospital's pregnancy training school will be planned. Birth Self-Efficacy Increasing Training Program Based on Motivational Interviewing Method for Pregnant Women 20-34. A four-session training program will be implemented, once a week for four weeks between weeks.

Control Group Within the scope of the research, no intervention will be made to the pregnant women in the control group between the 20th and 34th weeks, apart from the routine hospital practices.

Analysis of Research Data The descriptive statistics for the quantitative variables of the research determined by measurement will be shown as mean and standard deviation and percentage. First of all, the conformity of the data to the normal distribution will be evaluated with the Shapiro-Wilk test. In the analysis of normally distributed data as a result of the Shapiro-Wilk test, ANOVA between three or more variables and t-test in independent groups in pairwise comparisons, Mann-Whitney U test in pairwise comparisons between two-category variables in the analysis of non-parametric data, and Kruskal-Wallis H-test in order to find the differences between variables with three or more categories. Correlation analysis will be performed to reveal the relationship between dependent variables. In addition, Wilcoxon test (significance test of difference between two spouses) will be used to test the difference in two different measurement times obtained from the same individuals. The difference between categorical variables will be evaluated with the Pearson chi-square test. A value of 0.05 will be accepted as the level of significance in the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Being at least a primary school graduate,
* Being between 20-34 weeks in the calculations made according to the last menstrual date or with USG data for pregnant women who do not know the last menstrual date,
* Having a fear of birth,
* Having a single and live pregnancy,
* Agreeing to participate in the research,
* Having no difficulty in communicating,
* Without infertility treatment,
* No contraindications for vaginal birth

Exclusion Criteria:

* Pregnant women with medical indications,
* Those with risky pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since there is a training program on pregnant women, female gender was preferred.
Enrollment: 90 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
The Childbirth Self-Efficacy Scale-Short Form (CBSEI-SF) | each participant pregnant will be evaluated for outcome measure for four weeks
  The short version of the Birth Self-Efficacy Scale consists of 32 items. This scale was developed to measure the self-efficacy level of pregnant women in labor. The validity and reliability of the scale in Turkish was conducted. The scale consists of two sub-dimensions: outcome expectation and competence expectation. Each sub-dimension of the scale consists of 16 items. A high score from each subscale indicates that pregnant women have high expectations of adequacy and outcome regarding labor. High scores from the scale indicate that pregnant women have high self-efficacy levels in labor.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Sarı, Nurse, Principal Investigator — Yozgat City Hospital
Locations (1):
- Yozgat City Hospital, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected and affecting the outcome of the study will be published
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Only the collected data will be shared for analysis.